CLINICAL TRIAL: NCT01713335
Title: Proteasis Evaluation in COPD
Acronym: Pro-BPCO
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C11-56; 2012-A00885-38 (Registry Identifier: IDRCB)
Record Dates: First submitted 2012-10-15; First posted 2012-10-24 (Estimated); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sputum
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study was to evaluate kallikreins and its substrate, CCN, in COPD patients. Kallikreins are a subgroup of serine proteases, enzymes which are able to cleave peptide bonds in proteins. Kallicrein profile is unkonwn in COPD. The investigators will assess Kallikrein 1 to 15 and CCN 1 to 6 in sputum of patients. Three groups of patients will be included: Healthy smoker subjects, stable COPD patients and COPD patients with acute exacerbation. Kallicrein levels in sputum will be compared in these groups.

ELIGIBILITY:
Inclusion Criteria for healthy subjects:

* Smoker with tobacco consumption of 20 pack/year
* Normal lung function tests

Exclusion Criteria for healthy subjects:

* diagnosis of lung disease during the study
* Asthma
* Lung cancer
* Pregnant and lactating women

Inclusion Criteria for stable COPD:

* Smoker with tobacco consumption of 20 pack/year
* FEV1/FVC<70% on lung function tests
* no hospitalisation for exacerbation during 3 months before inclusion

Exclusion Criteria for stable COPD:

* Asthma
* Lung cancer
* Pregnant and lactating women

Inclusion Criteria for COPD with exacerbation:

* Smoker with tobacco consumption of 20 pack/year
* worsening of pulmonary symptoms
* FEV1/FVC<70% on lung function tests could be obtain before or 3 months after exacerbation

Exclusion Criteria for COPD with exacerbation:

* Asthma
* Lung cancer
* Pregnant and lactating women

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stable COPD patients were recruited from pulmonary primary care of pulmonary division of CHRU of Tours.
  COPD with acute exacerbation were recruited from hospitalisation of pulmonary division of CHRU of Tours and intensive care unit of CHRU of Tours.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2012-10-18 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Kallikrein level in sputum by ELISA | One sample at inclusion

SECONDARY OUTCOMES:
Comparison between kallikrein level and clinical or functionnal parameters | All data will be identified at inclusion
  Correlation between kallikrein and FEV1 Correlation between kallikrein and dyspnea score

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Guilleminault, MD, Principal Investigator — Service de Pneumologie, CHRU Tours, Tours, France; Valérie Gissot, MD, Principal Investigator — Centre d'Investigation Clinique, CHRU Tours, Tours, France; Antoine Guillon, MD, Principal Investigator — Service de Réanimation médicale, CHRU Tours, Tours, France
Locations (1):
- CHRU Tours, Tours, France